CLINICAL TRIAL: NCT06935110
Title: Feasibility of Tracheobronchial Defect Reconstruction Using Allogenic Aortic Patch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202407061DINE
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-04

CONDITIONS: Trachea Diseases; Airway Remodeling; Reconstruction Surgery
Keywords: cryopreserved aortic patch; airway repair; tracheal reconstruction; bronchial reconstruction
MeSH Terms: conditions — Tracheal Diseases; Airway Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryopreserved aortic patch (Experimental): Using the cryopreserve aortic patch to repair the tracheobronchial defect.
  Interventions: Procedure: Cryopreserved aortic patch

INTERVENTIONS:
Procedure: Cryopreserved aortic patch — After identifying the tracheal or bronchial defect with standard surgical techniques, the airway gap is reconstructed with a patch of human cryopreserved (-80 celsius degree) aortic allograft, which was not matched by the ABO and leukocyte antigen systems. The anastomosis is performed with standard technique for airway anastomosis. An silicon stent is inserted to prevent collapse for the aortic graft.

SUMMARY:
The investigators investigate the feasibility and safety of using cryopreserved aortic patches for tracheal or bronchial defect repair.

ELIGIBILITY:
Inclusion Criteria:

1. Congenital tracheal deformities: Includes congenital tracheomalacia, congenital tracheobronchial malformations, complete tracheal rings, etc., with severe clinical symptoms and cases where treatment is recommended after evaluation.
2. Acquired tracheal stenosis: Includes tracheal narrowing caused by diseases, endotracheal intubation, or postoperative scar tissue, with severe clinical symptoms and cases where treatment is recommended after evaluation.
3. Tracheal injury or tissue defect caused by trauma or burns: Cases requiring surgical repair.
4. Tracheal tumors: Reconstruction of tracheal tissue following the removal of benign or malignant tumors.

Exclusion Criteria:

1. Patients who are unable to provide informed consent.
2. Pulmonary tumors that can be treated with standard lobectomy.
3. Locally invasive tumors that are unresectable.
4. Presence of contralateral lymph node metastasis.
5. Presence of distant metastasis, except for solitary, resectable brain metastasis.
6. Tracheal lesions amenable to standard resection with direct anastomosis.
7. Preoperative evaluation indicates inability to undergo standard lobectomy.
8. Patients infected with human immunodeficiency virus (HIV) or with other immunodeficiency disorders.
9. Any condition or circumstance deemed by the principal investigator to potentially interfere with the conduct of the trial (e.g., severely impaired cardiopulmonary function, significant liver or kidney dysfunction, poorly controlled diabetes, high-risk groups, or pregnancy).
10. Individuals with concerns about the potential risks of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days
  The rate of death at 90 days.

SECONDARY OUTCOMES:
90-day morbidity | 90 days
  The occurrence of complication including 1) anastomotic leakage, 2) pneumonia, 3) difficult weaning, 4) airway obstruction by granulation tissue, 5) stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital, Taipei, 100
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung WT, Liao HC, Hsu HH, Chen JS. Stented cryopreserved aortic allograft for reconstruction of long-segment post-tuberculosis tracheal stenosis. J Formos Med Assoc. 2024 Jul;123(7):818-820. doi: 10.1016/j.jfma.2024.03.006. Epub 2024 Mar 16. PMID 38494361
- [Background] Martinod E, Radu DM, Onorati I, Portela AMS, Peretti M, Guiraudet P, Destable MD, Uzunhan Y, Freynet O, Chouahnia K, Duchemann B, Kabbani J, Maurer C, Brillet PY, Fath L, Brenet E, Debry C, Buffet C, Leenhardt L, Clero D, Julien N, Venissac N, Tronc F, Dutau H, Marquette CH, Juvin C, Lebreton G, Cohen Y, Zogheib E, Beloucif S, Planes C, Tresallet C, Bensidhoum M, Petite H, Rouard H, Miyara M, Vicaut E. Airway replacement using stented aortic matrices: Long-term follow-up and results of the TRITON-01 study in 35 adult patients. Am J Transplant. 2022 Dec;22(12):2961-2970. doi: 10.1111/ajt.17137. Epub 2022 Jul 14. PMID 35778956
- [Background] Martinod E, Chouahnia K, Radu DM, Joudiou P, Uzunhan Y, Bensidhoum M, Santos Portela AM, Guiraudet P, Peretti M, Destable MD, Solis A, Benachi S, Fialaire-Legendre A, Rouard H, Collon T, Piquet J, Leroy S, Venissac N, Santini J, Tresallet C, Dutau H, Sebbane G, Cohen Y, Beloucif S, d'Audiffret AC, Petite H, Valeyre D, Carpentier A, Vicaut E. Feasibility of Bioengineered Tracheal and Bronchial Reconstruction Using Stented Aortic Matrices. JAMA. 2018 Jun 5;319(21):2212-2222. doi: 10.1001/jama.2018.4653. PMID 29800033
- [Background] Karkhanis T, Byju AG, Morales DL, Zafar F, Haridas B. Composite Biosynthetic Graft for Repair of Long-Segment Tracheal Stenosis: A Pilot In Vivo and In Vitro Feasibility Study. ASAIO J. 2024 Jun 1;70(6):527-534. doi: 10.1097/MAT.0000000000002130. Epub 2024 Jan 3. PMID 38170278
- [Background] Allen MS. Surgery of the Trachea. Korean J Thorac Cardiovasc Surg. 2015 Aug;48(4):231-7. doi: 10.5090/kjtcs.2015.48.4.231. Epub 2015 Aug 5. PMID 26290833
- [Background] Etienne H, Fabre D, Gomez Caro A, Kolb F, Mussot S, Mercier O, Mitilian D, Stephan F, Fadel E, Dartevelle P. Tracheal replacement. Eur Respir J. 2018 Feb 14;51(2):1702211. doi: 10.1183/13993003.02211-2017. Print 2018 Feb. PMID 29444919
- [Background] Grillo HC. Development of tracheal surgery: a historical review. Part 2: Treatment of tracheal diseases. Ann Thorac Surg. 2003 Mar;75(3):1039-47. doi: 10.1016/s0003-4975(02)04109-7. No abstract available. PMID 12645751
- [Background] Grillo HC. Development of tracheal surgery: a historical review. Part 1: Techniques of tracheal surgery. Ann Thorac Surg. 2003 Feb;75(2):610-9. doi: 10.1016/s0003-4975(02)04108-5. No abstract available. PMID 12607695
- [Background] Madden BP. Evolutional trends in the management of tracheal and bronchial injuries. J Thorac Dis. 2017 Jan;9(1):E67-E70. doi: 10.21037/jtd.2017.01.43. PMID 28203439
- [Background] Prokakis C, Koletsis EN, Dedeilias P, Fligou F, Filos K, Dougenis D. Airway trauma: a review on epidemiology, mechanisms of injury, diagnosis and treatment. J Cardiothorac Surg. 2014 Jun 30;9:117. doi: 10.1186/1749-8090-9-117. PMID 24980209